CLINICAL TRIAL: NCT00552669
Title: Phase 4 Study of Randomized Comparison Among Oral Rapamycin Plus Bare Metal Stents Versus Drug Eluting Stents in de Novo Coronary Lesions.
Brief Title: Study of Oral Rapamycin Plus Bare Metal Stents vs Drug Eltuting Stents
Acronym: ORAR III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de estudios en Cardiologia Intervencionista (Other)
Responsible Party: Alfredo E Rodriguez, MD, PHD, FACC, FSCAI, Centro de Estudios en Cardiologia Intervencionista
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-Rodriguez; 01-CECI (Other: Sanatorio Otamendi y Miroli, Buenos Aires, Argentina); 02-IMA (Other: Clinica IMA, Buenos Aires, Argentina)
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Results first posted 2009-08-20 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Heart Disease; Coronary Restenosis
Keywords: Drug Eluting Stents; Stents Bare Metal; Stent Thrombosis; Coronary revascularization; Survival
MeSH Terms: conditions — Coronary Disease; Coronary Restenosis | interventions — Sirolimus; Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A--Oral Rapamycin plus BMS (Experimental): Oral sirolimus plus bare metal stent implantation
  Interventions: Drug: Oral sirolimus
- B -- Drug Eluting Stent (Active Comparator): Drug Eluting Stents
  Interventions: Device: Drug Eluting stent

INTERVENTIONS:
Drug: Oral sirolimus — Oral sirolimus given orally during 14 days plus bare metal stent implantation was compared with DES.Oral sirolimus was given as bolus of 10 mg started day before intervention followed by 3mg per day during 13 days after PCI. 180 mg of Diltiazem was added during oral administration of sirolimus .
  Other Names: Oral rapamycine
  Arms: A--Oral Rapamycin plus BMS
Device: Drug Eluting stent — Any Drug eluting stent
  Other Names: DES=Drug Eluting Stents); PES (Paclitaxel Eluting Stent); SES (Sirolimus eluting stent); ZES (Zotarolimus eluting stent)
  Arms: B -- Drug Eluting Stent

SUMMARY:
In a previous randomized comparison oral sirolimus plus bare metal stent compared to bare metal stent implantation alone demonstrated at one year of follow up a significant reduction of angiographic and clinical parameters of restenosis (ANMAT resolution number 3366 from June 2004 and Rodriguez A et al JACC,2006,47,1522-1529). In addition previous reported registries from our group with Drug Eluting Stents showed similar amount of reduction in clinical parameters (not angiographic)of restenosis (ERACI III, Rodriguez A et al EuroIntervention 2006,2:53-60). Taking in account that 8.3% of patients treated with oral rapamycin plus Bare Metal Stents(ORAR II Trial JACC 2006)and 8.8% of patients treated with DES developed clinical restenosis (ERACI III Registry, EuroIntervention 2006) the investigators sought to compare differences in overall cost with both revascularization strategies at 1, 2, 3 and 5 years of follow up assuming that safety and efficacy clinical end points would be similar.

DETAILED DESCRIPTION:
Patients with de novo lesions treated in different Institutions in Buenos Aires Argentina were randomized to treat with oral sirolimus plus bare metal stent implantation (100 patients) or DES(100 patients).

ELIGIBILITY:
Inclusion Criteria:

* Indication of revascularization
* De novo lesions
* Native vessels
* Suitable for stent placement

Exclusion Criteria:

* Acute myocardial infarction within the last 24 hours
* In stent restenosis
* Previous percutaneous coronary intervention within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo E Rodriguez, MD PhD FACC, Study Chair — Departamento de Cardiologia Intervencionista, Sanatorio Otamendi; Carlos Fernandez Pereira, MD, Study Director — Departamento de Cardiologia Intervencionista, Sanatorio Otamendi
Locations (3):
- Argentina (3):
  - Clinica IMA, Adrogué, Buenos Aires
  - Sanatorio Otamendi y Miroli, Buenos Aires, Buenos Aires
  - Sanatorio Las Lomas, San Isidro, Buenos Aires

REFERENCES:
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Schofer J, Schluter M, Gershlick AH, Wijns W, Garcia E, Schampaert E, Breithardt G; E-SIRIUS Investigators. Sirolimus-eluting stents for treatment of patients with long atherosclerotic lesions in small coronary arteries: double-blind, randomised controlled trial (E-SIRIUS). Lancet. 2003 Oct 4;362(9390):1093-9. doi: 10.1016/S0140-6736(03)14462-5. PMID 14550694
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Colombo A, Drzewiecki J, Banning A, Grube E, Hauptmann K, Silber S, Dudek D, Fort S, Schiele F, Zmudka K, Guagliumi G, Russell ME; TAXUS II Study Group. Randomized study to assess the effectiveness of slow- and moderate-release polymer-based paclitaxel-eluting stents for coronary artery lesions. Circulation. 2003 Aug 19;108(7):788-94. doi: 10.1161/01.CIR.0000086926.62288.A6. Epub 2003 Aug 4. PMID 12900339
- [Background] Virmani R, Guagliumi G, Farb A, Musumeci G, Grieco N, Motta T, Mihalcsik L, Tespili M, Valsecchi O, Kolodgie FD. Localized hypersensitivity and late coronary thrombosis secondary to a sirolimus-eluting stent: should we be cautious? Circulation. 2004 Feb 17;109(6):701-5. doi: 10.1161/01.CIR.0000116202.41966.D4. Epub 2004 Jan 26. PMID 14744976
- [Background] Pfisterer M, Brunner-La Rocca HP, Buser PT, Rickenbacher P, Hunziker P, Mueller C, Jeger R, Bader F, Osswald S, Kaiser C; BASKET-LATE Investigators. Late clinical events after clopidogrel discontinuation may limit the benefit of drug-eluting stents: an observational study of drug-eluting versus bare-metal stents. J Am Coll Cardiol. 2006 Dec 19;48(12):2584-91. doi: 10.1016/j.jacc.2006.10.026. Epub 2006 Nov 2. PMID 17174201
- [Background] Spaulding C, Daemen J, Boersma E, Cutlip DE, Serruys PW. A pooled analysis of data comparing sirolimus-eluting stents with bare-metal stents. N Engl J Med. 2007 Mar 8;356(10):989-97. doi: 10.1056/NEJMoa066633. Epub 2007 Feb 12. PMID 17296825
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Rodriguez AE, Mieres J, Fernandez-Pereira C, Vigo CF, Rodriguez-Alemparte M, Berrocal D, Grinfeld L, Palacios I. Coronary stent thrombosis in the current drug-eluting stent era: insights from the ERACI III trial. J Am Coll Cardiol. 2006 Jan 3;47(1):205-7. doi: 10.1016/j.jacc.2005.10.016. Epub 2005 Dec 9. No abstract available. PMID 16386687
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Hofma SH, van der Giessen WJ, van Dalen BM, Lemos PA, McFadden EP, Sianos G, Ligthart JM, van Essen D, de Feyter PJ, Serruys PW. Indication of long-term endothelial dysfunction after sirolimus-eluting stent implantation. Eur Heart J. 2006 Jan;27(2):166-70. doi: 10.1093/eurheartj/ehi571. Epub 2005 Oct 25. PMID 16249221
- [Background] Gallo R, Padurean A, Jayaraman T, Marx S, Roque M, Adelman S, Chesebro J, Fallon J, Fuster V, Marks A, Badimon JJ. Inhibition of intimal thickening after balloon angioplasty in porcine coronary arteries by targeting regulators of the cell cycle. Circulation. 1999 Apr 27;99(16):2164-70. doi: 10.1161/01.cir.99.16.2164. PMID 10217658
- [Background] Poon M, Marx SO, Gallo R, Badimon JJ, Taubman MB, Marks AR. Rapamycin inhibits vascular smooth muscle cell migration. J Clin Invest. 1996 Nov 15;98(10):2277-83. doi: 10.1172/JCI119038. PMID 8941644
- [Background] Rodriguez AE, Alemparte MR, Vigo CF, Pereira CF, Llaurado C, Russo M, Virmani R, Ambrose JA. Pilot study of oral rapamycin to prevent restenosis in patients undergoing coronary stent therapy: Argentina Single-Center Study (ORAR Trial). J Invasive Cardiol. 2003 Oct;15(10):581-4. PMID 14519892
- [Background] Hausleiter J, Kastrati A, Mehilli J, Vogeser M, Zohlnhofer D, Schuhlen H, Goos C, Pache J, Dotzer F, Pogatsa-Murray G, Dirschinger J, Heemann U, Schomig A; OSIRIS Investigators. Randomized, double-blind, placebo-controlled trial of oral sirolimus for restenosis prevention in patients with in-stent restenosis: the Oral Sirolimus to Inhibit Recurrent In-stent Stenosis (OSIRIS) trial. Circulation. 2004 Aug 17;110(7):790-5. doi: 10.1161/01.CIR.0000138935.17503.35. Epub 2004 Aug 9. PMID 15302787
- [Background] Waksman R, Ajani AE, Pichard AD, Torguson R, Pinnow E, Canos D, Satler LF, Kent KM, Kuchulakanti P, Pappas C, Gambone L, Weissman N, Abbott MC, Lindsay J; Oral Rapamune to Inhibit Restenosis study. Oral rapamycin to inhibit restenosis after stenting of de novo coronary lesions: the Oral Rapamune to Inhibit Restenosis (ORBIT) study. J Am Coll Cardiol. 2004 Oct 6;44(7):1386-92. doi: 10.1016/j.jacc.2004.06.069. PMID 15464317
- [Background] Rodriguez AE, Rodriguez Alemparte M, Vigo CF, Fernandez Pereira C, Llaurado C, Vetcher D, Pocovi A, Ambrose J. Role of oral rapamycin to prevent restenosis in patients with de novo lesions undergoing coronary stenting: results of the Argentina single centre study (ORAR trial). Heart. 2005 Nov;91(11):1433-7. doi: 10.1136/hrt.2004.050617. Epub 2005 Mar 17. PMID 15774608
- [Background] Rodriguez AE, Granada JF, Rodriguez-Alemparte M, Vigo CF, Delgado J, Fernandez-Pereira C, Pocovi A, Rodriguez-Granillo AM, Schulz D, Raizner AE, Palacios I, O'Neill W, Kaluza GL, Stone G; ORAR II Investigators. Oral rapamycin after coronary bare-metal stent implantation to prevent restenosis: the Prospective, Randomized Oral Rapamycin in Argentina (ORAR II) Study. J Am Coll Cardiol. 2006 Apr 18;47(8):1522-9. doi: 10.1016/j.jacc.2005.12.052. Epub 2006 Mar 29. PMID 16630986
- [Background] Stone GW, Ellis SG, Cannon L, Mann JT, Greenberg JD, Spriggs D, O'Shaughnessy CD, DeMaio S, Hall P, Popma JJ, Koglin J, Russell ME; TAXUS V Investigators. Comparison of a polymer-based paclitaxel-eluting stent with a bare metal stent in patients with complex coronary artery disease: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1215-23. doi: 10.1001/jama.294.10.1215. PMID 16160130
- [Background] Beohar N, Davidson CJ, Kip KE, Goodreau L, Vlachos HA, Meyers SN, Benzuly KH, Flaherty JD, Ricciardi MJ, Bennett CL, Williams DO. Outcomes and complications associated with off-label and untested use of drug-eluting stents. JAMA. 2007 May 9;297(18):1992-2000. doi: 10.1001/jama.297.18.1992. PMID 17488964
- [Background] Win HK, Caldera AE, Maresh K, Lopez J, Rihal CS, Parikh MA, Granada JF, Marulkar S, Nassif D, Cohen DJ, Kleiman NS; EVENT Registry Investigators. Clinical outcomes and stent thrombosis following off-label use of drug-eluting stents. JAMA. 2007 May 9;297(18):2001-9. doi: 10.1001/jama.297.18.2001. PMID 17488965
- [Background] Rodriguez AE, Maree AO, Mieres J, Berrocal D, Grinfeld L, Fernandez-Pereira C, Curotto V, Rodriguez-Granillo A, O'Neill W, Palacios IF. Late loss of early benefit from drug-eluting stents when compared with bare-metal stents and coronary artery bypass surgery: 3 years follow-up of the ERACI III registry. Eur Heart J. 2007 Sep;28(17):2118-25. doi: 10.1093/eurheartj/ehm297. Epub 2007 Jul 25. PMID 17656352
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Morice MC, Colombo A, Meier B, Serruys P, Tamburino C, Guagliumi G, Sousa E, Stoll HP; REALITY Trial Investigators. Sirolimus- vs paclitaxel-eluting stents in de novo coronary artery lesions: the REALITY trial: a randomized controlled trial. JAMA. 2006 Feb 22;295(8):895-904. doi: 10.1001/jama.295.8.895. PMID 16493102
- [Background] Kandzari DE, Leon MB, Popma JJ, Fitzgerald PJ, O'Shaughnessy C, Ball MW, Turco M, Applegate RJ, Gurbel PA, Midei MG, Badre SS, Mauri L, Thompson KP, LeNarz LA, Kuntz RE; ENDEAVOR III Investigators. Comparison of zotarolimus-eluting and sirolimus-eluting stents in patients with native coronary artery disease: a randomized controlled trial. J Am Coll Cardiol. 2006 Dec 19;48(12):2440-7. doi: 10.1016/j.jacc.2006.08.035. Epub 2006 Nov 28. PMID 17174180
- [Background] Agostoni P, Valgimigli M, Abbate A, Cosgrave J, Pilati M, Biondi-Zoccai GG. Is late luminal loss an accurate predictor of the clinical effectiveness of drug-eluting stents in the coronary arteries? Am J Cardiol. 2006 Mar 1;97(5):603-5. doi: 10.1016/j.amjcard.2005.09.095. Epub 2006 Jan 6. PMID 16490421
- [Background] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Background] Togni M, Windecker S, Cocchia R, Wenaweser P, Cook S, Billinger M, Meier B, Hess OM. Sirolimus-eluting stents associated with paradoxic coronary vasoconstriction. J Am Coll Cardiol. 2005 Jul 19;46(2):231-6. doi: 10.1016/j.jacc.2005.01.062. PMID 16022947
- [Background] Kotani J, Awata M, Nanto S, Uematsu M, Oshima F, Minamiguchi H, Mintz GS, Nagata S. Incomplete neointimal coverage of sirolimus-eluting stents: angioscopic findings. J Am Coll Cardiol. 2006 May 16;47(10):2108-11. doi: 10.1016/j.jacc.2005.11.092. Epub 2006 Apr 4. PMID 16697331
- [Background] Spertus JA, Kettelkamp R, Vance C, Decker C, Jones PG, Rumsfeld JS, Messenger JC, Khanal S, Peterson ED, Bach RG, Krumholz HM, Cohen DJ. Prevalence, predictors, and outcomes of premature discontinuation of thienopyridine therapy after drug-eluting stent placement: results from the PREMIER registry. Circulation. 2006 Jun 20;113(24):2803-9. doi: 10.1161/CIRCULATIONAHA.106.618066. Epub 2006 Jun 12. PMID 16769908
- [Background] Buonamici P, Marcucci R, Migliorini A, Gensini GF, Santini A, Paniccia R, Moschi G, Gori AM, Abbate R, Antoniucci D. Impact of platelet reactivity after clopidogrel administration on drug-eluting stent thrombosis. J Am Coll Cardiol. 2007 Jun 19;49(24):2312-7. doi: 10.1016/j.jacc.2007.01.094. Epub 2007 Jun 4. PMID 17572245
- [Background] Ho PM, Peterson ED, Wang L, Magid DJ, Fihn SD, Larsen GC, Jesse RA, Rumsfeld JS. Incidence of death and acute myocardial infarction associated with stopping clopidogrel after acute coronary syndrome. JAMA. 2008 Feb 6;299(5):532-9. doi: 10.1001/jama.299.5.532. PMID 18252883
- [Background] Brunner-La Rocca HP, Kaiser C, Bernheim A, Zellweger MJ, Jeger R, Buser PT, Osswald S, Pfisterer M; BASKET Investigators. Cost-effectiveness of drug-eluting stents in patients at high or low risk of major cardiac events in the Basel Stent KostenEffektivitats Trial (BASKET): an 18-month analysis. Lancet. 2007 Nov 3;370(9598):1552-9. doi: 10.1016/S0140-6736(07)61660-2. PMID 17980734
- [Background] Cohen DJ, Bakhai A, Shi C, Githiora L, Lavelle T, Berezin RH, Leon MB, Moses JW, Carrozza JP Jr, Zidar JP, Kuntz RE; SIRIUS Investigators. Cost-effectiveness of sirolimus-eluting stents for treatment of complex coronary stenoses: results from the Sirolimus-Eluting Balloon Expandable Stent in the Treatment of Patients With De Novo Native Coronary Artery Lesions (SIRIUS) trial. Circulation. 2004 Aug 3;110(5):508-14. doi: 10.1161/01.CIR.0000136821.99814.43. Epub 2004 Jul 19. PMID 15262844
- [Background] Bakhai A, Stone GW, Mahoney E, Lavelle TA, Shi C, Berezin RH, Lahue BJ, Clark MA, Lacey MJ, Russell ME, Ellis SG, Hermiller JB, Cox DA, Cohen DJ; TAXUS-IV Investigators. Cost effectiveness of paclitaxel-eluting stents for patients undergoing percutaneous coronary revascularization: results from the TAXUS-IV Trial. J Am Coll Cardiol. 2006 Jul 18;48(2):253-61. doi: 10.1016/j.jacc.2006.02.063. Epub 2006 Jun 22. PMID 16843171
- [Background] Hausleiter J, Kastrati A. Is there a role for oral rapamycin in restenosis prevention after bare-metal stent implantation? Nat Clin Pract Cardiovasc Med. 2006 Sep;3(9):476-7. doi: 10.1038/ncpcardio0633. No abstract available. PMID 16932762
- [Derived] Rodriguez AE, Rodriguez-Granillo AM, Antoniucci D, Mieres J, Fernandez-Pereira C, Rodriguez-Granillo GA, Santaera O, Rubilar B, Palacios IF, Serruys PW; ORAR III Investigators. Randomized comparison of cost-saving and effectiveness of oral rapamycin plus bare-metal stents with drug-eluting stents: three-year outcome from the randomized oral rapamycin in Argentina (ORAR) III trial. Catheter Cardiovasc Interv. 2012 Sep 1;80(3):385-94. doi: 10.1002/ccd.23352. Epub 2011 Dec 8. PMID 22109997
- [Derived] Rodriguez AE, Maree A, Tarragona S, Fernandez-Pereira C, Santaera O, Rodriguez Granillo AM, Rodriguez-Granillo GA, Russo-Felssen M, Kukreja N, Antoniucci D, Palacios IF, Serruys PW; ORAR III Investigators. Percutaneous coronary intervention with oral sirolimus and bare metal stents has comparable safety and efficacy to treatment with drug eluting stents, but with significant cost saving: long-term follow-up results from the randomised, controlled ORAR III (Oral Rapamycin in ARgentina) study. EuroIntervention. 2009 Jun;5(2):255-64. doi: 10.4244/eijv5i2a40. PMID 20449934
- See also: Pubmed abstract of the latest published results. — http://www.ncbi.nlm.nih.gov/sites/entrez

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2006 to September 2007 we enrolled 200 patients in the trial.
Pre-assignment Details: From 1274 patients with coronary angiography, 789 met clinical inclusion criteria, from whom 102 have angiographic exclusion criteria. 487 were excluded for inability for percutaneous coronary intervention (PCI) with drug eluting stent (DES) deployment or refuse to participate in the study; thus 200 patients were included in this randomized trial.
Groups:
- Oral Sirolimus + Bare Metal Stent: Oral sirolimus plus bare metal stent implantation
- Drug Eluting Stents: Any Drug Eluting Stents
Period: Overall Study
Arm/Group | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents
Started | 100 (patients) | 100 (patients)
Completed | 97 (All patients were followed for 18.3 +/- 7 months.) | 93 (All patients were followed for 18.3 +/- 7 months.)
Not Completed | 3 | 7
Not completed — Death | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 58 | 119
  >=65 years | 39 | 42 | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.1) | 63.4 (10.6) | 63.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 83 | 81 | 164
Region of Enrollment [Number; unit: participants]
  Argentina | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Differences in Costs Between Two Revascularization Strategies for de Novo Coronary Lesions.
Description: Overall costs expressed in US dollars at 18 months of follow up between Oral Sirolimus Plus BMS vs DES implantation in denovo coronary lesions.
Time Frame: Follow up will be conducted by the coordinating Center at 18 months of follow up
Population: All patients were analyzed for ITT and the imputation technique was LOCF
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents
Number analyzed (Participants) | 100 | 100
US dollars | 5483 (2165.5) | 7658.2 (3263.4)
Statistical Analysis 1: Comparison: Oral Sirolimus + Bare Metal Stent vs Drug Eluting Stents; We used One way annalysis of a variance for means and standard deviation; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Major Adverse Cardiovascular Events (MACCE)
Description: Death from any cause, myocardial infarction and stroke. Safety was analyzed as MACCE (major adverse cardiovascular events) including death, MI and stroke.
Time Frame: 18 Months
Population: It was determinated by ITT and the technique used was LOCF.
Measure: Number; unit: participants
Arm/Group | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents
Number analyzed (Participants) | 100 | 100
participants
  MACCE | 9 | 15
  Death | 3 | 7
  Acute Myocardial Infarction | 6 | 9
  Stroke | 0 | 1
Statistical Analysis 1: Comparison: Oral Sirolimus + Bare Metal Stent vs Drug Eluting Stents; Based on our previous data the incidence of relevant clinical events was similar in both groups (ERACI III and ORAR II); Test type: Superiority or Other; p = 0.05, Chi-squared

3. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: Efficacy end point was TVR as revasacularization of the treated vessel.
Time Frame: 18 months
Population: We analyzed the number of vessels treated per group by ITT and the imputation technique was LOCF.
Measure: Number; unit: vessels
Arm/Group | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents
Number analyzed (Participants) | 131 | 142
vessels | 14 | 15
Statistical Analysis 1: Comparison: Oral Sirolimus + Bare Metal Stent vs Drug Eluting Stents; power calculation 80% Hypothesis: No significant diferences between Target Vessel Revascularization (TVR) between both groups. All events will be recorded and an independent blind for groups clinical events committee will adjudicate each one; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents
Serious Adverse Events (participants affected / at risk) | 9 | 15
Other Adverse Events (participants affected / at risk) | 9/100 | 2/100
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Oral Sirolimus + Bare Metal Stent | Drug Eluting Stents
Acute Myocardial Infarction (Cardiac disorders) | 6/100 (9) | 9/100 (15)
Cardiac Death (Cardiac disorders) | 1/100 (9) | 4/100 (15)
Non Cardiac Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/100 (9) | 3/100 (15)
Stroke (Vascular disorders) | 0/100 (9) | 1/100 (15)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Sirolimus + Bare Metal Stent (N=100) | Drug Eluting Stents (N=100)
Allergy (Immune system disorders) | 3 (9) | 2 (2) — None hospitalization was needed for any participant patient
diarrhea (Gastrointestinal disorders) | 6 (9) | 0 (2) — None hospitalization was needed for any participant patient

LIMITATIONS AND CAVEATS:
It was an open label design. Multiple approved DES designs were used. Health Care system in Argentina differs from other world ones.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No